CLINICAL TRIAL: NCT02734238
Title: Physiological and Psychological Effects of Testosterone During Severe Energy Deficit and Recovery: a Randomized, Placebo Controlled Trial
Brief Title: Physiological and Psychological Effects of Testosterone During Severe Energy Deficit and Recovery
Acronym: OPS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency); MyoSyntax (Unknown); Defence Research and Development Canada (Industry); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jennifer C. Rood, Principal Investigator, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PBRC 2015-063
Record Dates: First submitted 2016-03-31; First posted 2016-04-12 (Estimated); Results first posted 2019-01-02 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Caloric Restriction; Exercise
MeSH Terms: conditions — Motor Activity | interventions — Sesame Oil; testosterone enanthate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Energy Deficit (Placebo Comparator): Participants randomly assigned to the control condition will be subject to exercise-induced energy expenditure resulting in a 55% energy deficit and will be administered sesame oil placebo injections during phase 2 of the trial.
  Interventions: Drug: Sesame Oil
- Energy Deficit + Testosterone (Experimental): Participants randomly assigned to the intervention condition will be subject to exercise-induced energy expenditure resulting in a 55% energy deficit and will be administered testosterone enanthate injections during phase 2 of the trial.
  Interventions: Drug: testosterone enanthate

INTERVENTIONS:
Drug: Sesame Oil — 200 mg sesame oil by intramuscular injection weekly on days 15, 21, 28, and 35
  Arms: Energy Deficit
Drug: testosterone enanthate — 200 mg testosterone enanthate by intramuscular injection weekly on days 15, 21, 28, and 35
  Arms: Energy Deficit + Testosterone

SUMMARY:
The objective of this study is to determine whether maintaining a eugonadal state, during severe, sustained energy deficit, attenuates physiological decrements, particularly the loss of lean body mass.

DETAILED DESCRIPTION:
This study will enroll up to 60 physically active men in a 3-phase randomized, placebo-controlled trial. After completing a 14-day (free-living, phase 1), energy-adequate, diet-acclimation phase (protein, 1.6 g∙kg-1∙d-1; fat 30% total energy intake, with remaining energy derived from carbohydrate), participants will be randomized to one of two experimental groups and undergo a 28-day (live-in, phase 2), 55% energy deficit phase: energy deficit alone (DEF) or energy deficit + exogenous testosterone (DEF+TEST). Recovery (free-living, phase 3) will be assessed after completing phase 2 to determine when body mass has been recovered within ± 2.5% of initial body mass (duration will vary, 42-day maximum for phase 3). This study will delineate the contribution of testosterone declines from the physical and mental demands encountered by Warfighters during military training and combat operations on complex markers of physiological and psychological status, addressing a direct, consistently observed, gap in knowledge.

ELIGIBILITY:
Inclusion Criteria:

* Physically active (at least 2 days per week aerobic and/or resistance exercise)
* Not taking any prescription medications and/or willing to refrain from all medication use prior to and throughout the entire study period, unless provided/approved by the study physician
* Willing to refrain from alcohol, smoking, e-cigarettes, or use of any nicotine product, caffeine, and dietary supplement use throughout the entire study period

  * At the discretion of the study physician, wash-out period for medications, supplements, and over-the-counter medications is ≥ 1 to 4 weeks
  * Wash-out period for caffeine and alcohol is ≥ 7 days
* Willing to live on the Pennington Biomedical Research Center inpatient unit for 28 consecutive days
* Willing to have a urine drug screening
* Meets age-specific U.S. Army body composition standards according to Army Regulation 600-9, which includes estimates of percent body fat based on height, weight, and circumference measures (neck and waist)
* Total testosterone concentration is within the normal physiological range, total testosterone (300-1,000 ng/dL).

Exclusion Criteria:

* Musculoskeletal injuries that compromise exercise capability
* Diagnosed cardiometabolic disorders (i.e., hypertension, hyperlipidemia, kidney disease, diabetes, etc.)
* Allergies or intolerance to foods, vegetarian practices, or history of complications with lidocaine
* Anabolic steroid, human growth hormone, or nutritional testosterone precursor-like supplement use within the past 6 months
* Will not refrain from smoking (any nicotine product), alcohol, caffeine, or any other dietary supplement during the study
* Any use of antibiotics, except topical antibiotics, within 3 months of study participation
* Colonoscopy within 3 months of study participation
* Chronic use of laxatives, stool softeners, antacids, or anti-diarrheal medications (≥ once a week)
* History of gastrointestinal disease (e.g., celiac, irritable bowel syndrome, colitis, Crohn's disease)
* Restrained eater (the Three-Factor Eating Questionnaire) as assessed by the study's psychological and behavioral assessment staff
* Adults unable to consent
* Women
* Prisoners
* Metal implants, claustrophobia, head size incompatible with MRI equipment, etc.
* Sedentary or engages in <2 days of physical activity per week (aerobic and/or resistance training)
* Exceeds age-specific U.S. Army body composition standards according to Army Regulation 600-9
* Previous history of kidney stones unless otherwise approved by the medical investigator
* Systolic blood pressure > 150 or diastolic blood pressure > 95 mmHg
* Previous history of breast or prostate cancer
* Previous history of Chronic Obstructive Pulmonary Disease or Obstructive Sleep Apnea
* Findings of lab results of prostate-specific antigen > 3ng/ml, Hematocrit > 50%, or positive urine drug screening
* Based on the investigative team's clinical judgment, a subject may not be appropriate for participation in the study

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer C Rood, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pasiakos SM, Margolis LM, Orr JS. Optimized dietary strategies to protect skeletal muscle mass during periods of unavoidable energy deficit. FASEB J. 2015 Apr;29(4):1136-42. doi: 10.1096/fj.14-266890. Epub 2014 Dec 30. PMID 25550460
- [Background] Lieberman HR, Thompson LA, Caruso CM, Niro PJ, Mahoney CR, McClung JP, Caron GR. The catecholamine neurotransmitter precursor tyrosine increases anger during exposure to severe psychological stress. Psychopharmacology (Berl). 2015 Mar;232(5):943-51. doi: 10.1007/s00213-014-3727-7. Epub 2014 Sep 16. PMID 25220844
- [Background] Friedl KE, Moore RJ, Hoyt RW, Marchitelli LJ, Martinez-Lopez LE, Askew EW. Endocrine markers of semistarvation in healthy lean men in a multistressor environment. J Appl Physiol (1985). 2000 May;88(5):1820-30. doi: 10.1152/jappl.2000.88.5.1820. PMID 10797147
- [Background] Opstad PK. The hypothalamo-pituitary regulation of androgen secretion in young men after prolonged physical stress combined with energy and sleep deprivation. Acta Endocrinol (Copenh). 1992 Sep;127(3):231-6. doi: 10.1530/acta.0.1270231. PMID 1414148
- [Background] Henning PC, Scofield DE, Spiering BA, Staab JS, Matheny RW Jr, Smith MA, Bhasin S, Nindl BC. Recovery of endocrine and inflammatory mediators following an extended energy deficit. J Clin Endocrinol Metab. 2014 Mar;99(3):956-64. doi: 10.1210/jc.2013-3046. Epub 2013 Dec 11. PMID 24423293
- [Background] Nindl BC, Friedl KE, Frykman PN, Marchitelli LJ, Shippee RL, Patton JF. Physical performance and metabolic recovery among lean, healthy men following a prolonged energy deficit. Int J Sports Med. 1997 Jul;18(5):317-24. doi: 10.1055/s-2007-972640. PMID 9298770
- [Background] Nindl BC, Alemany JA, Kellogg MD, Rood J, Allison SA, Young AJ, Montain SJ. Utility of circulating IGF-I as a biomarker for assessing body composition changes in men during periods of high physical activity superimposed upon energy and sleep restriction. J Appl Physiol (1985). 2007 Jul;103(1):340-6. doi: 10.1152/japplphysiol.01321.2006. Epub 2007 Apr 5. PMID 17412783
- [Background] Carbone JW, McClung JP, Pasiakos SM. Skeletal muscle responses to negative energy balance: effects of dietary protein. Adv Nutr. 2012 Mar 1;3(2):119-26. doi: 10.3945/an.111.001792. PMID 22516719
- [Background] Knapik JJ, Ang P, Meiselman H, Johnson W, Kirk J, Bensel C, Hanlon W. Soldier performance and strenuous road marching: influence of load mass and load distribution. Mil Med. 1997 Jan;162(1):62-7. PMID 9002707
- [Background] Knapik JJ, Reynolds KL, Harman E. Soldier load carriage: historical, physiological, biomechanical, and medical aspects. Mil Med. 2004 Jan;169(1):45-56. doi: 10.7205/milmed.169.1.45. PMID 14964502
- [Background] Roy TC. Diagnoses and mechanisms of musculoskeletal injuries in an infantry brigade combat team deployed to Afghanistan evaluated by the brigade physical therapist. Mil Med. 2011 Aug;176(8):903-8. doi: 10.7205/milmed-d-11-00006. PMID 21882780
- [Background] Roy TC, Ritland BM, Knapik JJ, Sharp MA. Lifting tasks are associated with injuries during the early portion of a deployment to Afghanistan. Mil Med. 2012 Jun;177(6):716-22. doi: 10.7205/milmed-d-11-00402. PMID 22730849
- [Background] Christensen PA, Jacobsen O, Thorlund JB, Madsen T, Moller C, Jensen C, Suetta C, Aagaard P. Changes in maximum muscle strength and rapid muscle force characteristics after long-term special support and reconnaissance missions: a preliminary report. Mil Med. 2008 Sep;173(9):889-94. doi: 10.7205/milmed.173.9.889. PMID 18816929
- [Background] Alemany JA, Nindl BC, Kellogg MD, Tharion WJ, Young AJ, Montain SJ. Effects of dietary protein content on IGF-I, testosterone, and body composition during 8 days of severe energy deficit and arduous physical activity. J Appl Physiol (1985). 2008 Jul;105(1):58-64. doi: 10.1152/japplphysiol.00005.2008. Epub 2008 May 1. PMID 18450989
- [Background] Hoyt RW, Opstad PK, Haugen AH, DeLany JP, Cymerman A, Friedl KE. Negative energy balance in male and female rangers: effects of 7 d of sustained exercise and food deprivation. Am J Clin Nutr. 2006 May;83(5):1068-75. doi: 10.1093/ajcn/83.5.1068. PMID 16685048
- [Background] Margolis LM, Rood J, Champagne C, Young AJ, Castellani JW. Energy balance and body composition during US Army special forces training. Appl Physiol Nutr Metab. 2013 Apr;38(4):396-400. doi: 10.1139/apnm-2012-0323. Epub 2013 Apr 3. PMID 23713532
- [Background] Nindl BC, Barnes BR, Alemany JA, Frykman PN, Shippee RL, Friedl KE. Physiological consequences of U.S. Army Ranger training. Med Sci Sports Exerc. 2007 Aug;39(8):1380-7. doi: 10.1249/MSS.0b013e318067e2f7. PMID 17762372
- [Background] Nindl BC, Rarick KR, Castellani JW, Tuckow AP, Patton JF, Young AJ, Montain SJ. Altered secretion of growth hormone and luteinizing hormone after 84 h of sustained physical exertion superimposed on caloric and sleep restriction. J Appl Physiol (1985). 2006 Jan;100(1):120-8. doi: 10.1152/japplphysiol.01415.2004. Epub 2005 Sep 1. PMID 16141374
- [Background] Nindl BC, Leone CD, Tharion WJ, Johnson RF, Castellani JW, Patton JF, Montain SJ. Physical performance responses during 72 h of military operational stress. Med Sci Sports Exerc. 2002 Nov;34(11):1814-22. doi: 10.1097/00005768-200211000-00019. PMID 12439088
- [Background] Welsh TT, Alemany JA, Montain SJ, Frykman PN, Tuckow AP, Young AJ, Nindl BC. Effects of intensified military field training on jumping performance. Int J Sports Med. 2008 Jan;29(1):45-52. doi: 10.1055/s-2007-964970. Epub 2007 Sep 18. PMID 17879876
- [Background] Thorlund JB, Jakobsen O, Madsen T, Christensen PA, Nedergaard A, Andersen JL, Suetta C, Aagaard P. Changes in muscle strength and morphology after muscle unloading in Special Forces missions. Scand J Med Sci Sports. 2011 Dec;21(6):e56-63. doi: 10.1111/j.1600-0838.2010.01149.x. Epub 2010 Jun 18. PMID 20561275
- [Background] Areta JL, Burke LM, Camera DM, West DW, Crawshay S, Moore DR, Stellingwerff T, Phillips SM, Hawley JA, Coffey VG. Reduced resting skeletal muscle protein synthesis is rescued by resistance exercise and protein ingestion following short-term energy deficit. Am J Physiol Endocrinol Metab. 2014 Apr 15;306(8):E989-97. doi: 10.1152/ajpendo.00590.2013. Epub 2014 Mar 4. PMID 24595305
- [Background] Wycherley TP, Moran LJ, Clifton PM, Noakes M, Brinkworth GD. Effects of energy-restricted high-protein, low-fat compared with standard-protein, low-fat diets: a meta-analysis of randomized controlled trials. Am J Clin Nutr. 2012 Dec;96(6):1281-98. doi: 10.3945/ajcn.112.044321. Epub 2012 Oct 24. PMID 23097268
- [Background] Pasiakos SM, Cao JJ, Margolis LM, Sauter ER, Whigham LD, McClung JP, Rood JC, Carbone JW, Combs GF Jr, Young AJ. Effects of high-protein diets on fat-free mass and muscle protein synthesis following weight loss: a randomized controlled trial. FASEB J. 2013 Sep;27(9):3837-47. doi: 10.1096/fj.13-230227. Epub 2013 Jun 5. PMID 23739654
- [Background] Pasiakos SM, Margolis LM, McClung JP, Cao JJ, Whigham LD, Combs GF, Young AJ. Whole-body protein turnover response to short-term high-protein diets during weight loss: a randomized controlled trial. Int J Obes (Lond). 2014 Jul;38(7):1015-8. doi: 10.1038/ijo.2013.197. Epub 2013 Oct 29. PMID 24166063
- [Background] Pasiakos SM, Austin KG, Lieberman HR, Askew EW. Efficacy and safety of protein supplements for U.S. Armed Forces personnel: consensus statement. J Nutr. 2013 Nov;143(11):1811S-1814S. doi: 10.3945/jn.113.176859. Epub 2013 Sep 11. PMID 24027189
- [Background] Margolis LM, Murphy NE, Martini S, Spitz MG, Thrane I, McGraw SM, Blatny JM, Castellani JW, Rood JC, Young AJ, Montain SJ, Gundersen Y, Pasiakos SM. Effects of winter military training on energy balance, whole-body protein balance, muscle damage, soreness, and physical performance. Appl Physiol Nutr Metab. 2014 Dec;39(12):1395-401. doi: 10.1139/apnm-2014-0212. PMID 25386980
- [Background] Bhasin S, Woodhouse L, Casaburi R, Singh AB, Bhasin D, Berman N, Chen X, Yarasheski KE, Magliano L, Dzekov C, Dzekov J, Bross R, Phillips J, Sinha-Hikim I, Shen R, Storer TW. Testosterone dose-response relationships in healthy young men. Am J Physiol Endocrinol Metab. 2001 Dec;281(6):E1172-81. doi: 10.1152/ajpendo.2001.281.6.E1172. PMID 11701431
- [Background] Finkelstein JS, Yu EW, Burnett-Bowie SA. Gonadal steroids and body composition, strength, and sexual function in men. N Engl J Med. 2013 Dec 19;369(25):2457. doi: 10.1056/NEJMc1313169. No abstract available. PMID 24350954
- [Background] Kvorning T, Andersen M, Brixen K, Madsen K. Suppression of endogenous testosterone production attenuates the response to strength training: a randomized, placebo-controlled, and blinded intervention study. Am J Physiol Endocrinol Metab. 2006 Dec;291(6):E1325-32. doi: 10.1152/ajpendo.00143.2006. Epub 2006 Jul 25. PMID 16868226
- [Background] Mauras N, Hayes V, Welch S, Rini A, Helgeson K, Dokler M, Veldhuis JD, Urban RJ. Testosterone deficiency in young men: marked alterations in whole body protein kinetics, strength, and adiposity. J Clin Endocrinol Metab. 1998 Jun;83(6):1886-92. doi: 10.1210/jcem.83.6.4892. PMID 9626114
- [Background] Henning PC, Margolis LM, McClung JP, Young AJ, Pasiakos SM. High protein diets do not attenuate decrements in testosterone and IGF-I during energy deficit. Metabolism. 2014 May;63(5):628-32. doi: 10.1016/j.metabol.2014.02.007. Epub 2014 Feb 17. PMID 24641883
- [Background] Murphy MG, Plunkett LM, Gertz BJ, He W, Wittreich J, Polvino WM, Clemmons DR. MK-677, an orally active growth hormone secretagogue, reverses diet-induced catabolism. J Clin Endocrinol Metab. 1998 Feb;83(2):320-5. doi: 10.1210/jcem.83.2.4551. PMID 9467534
- [Background] Clemmons DR, Smith-Banks A, Underwood LE. Reversal of diet-induced catabolism by infusion of recombinant insulin-like growth factor-I in humans. J Clin Endocrinol Metab. 1992 Jul;75(1):234-8. doi: 10.1210/jcem.75.1.1619015.
- [Background] Kupfer SR, Underwood LE, Baxter RC, Clemmons DR. Enhancement of the anabolic effects of growth hormone and insulin-like growth factor I by use of both agents simultaneously. J Clin Invest. 1993 Feb;91(2):391-6. doi: 10.1172/JCI116212. PMID 7679407
- [Background] Dulloo AG, Jacquet J, Montani JP. How dieting makes some fatter: from a perspective of human body composition autoregulation. Proc Nutr Soc. 2012 Aug;71(3):379-89. doi: 10.1017/S0029665112000225. Epub 2012 Apr 5. PMID 22475574
- [Background] Dulloo AG, Jacquet J, Girardier L. Poststarvation hyperphagia and body fat overshooting in humans: a role for feedback signals from lean and fat tissues. Am J Clin Nutr. 1997 Mar;65(3):717-23. doi: 10.1093/ajcn/65.3.717. PMID 9062520
- [Background] Pescatello LS, Devaney JM, Hubal MJ, Thompson PD, Hoffman EP. Highlights from the functional single nucleotide polymorphisms associated with human muscle size and strength or FAMuSS study. Biomed Res Int. 2013;2013:643575. doi: 10.1155/2013/643575. Epub 2013 Dec 23. PMID 24455711
- [Background] Silverman I, Kastuk D, Choi J, Phillips K. Testosterone levels and spatial ability in men. Psychoneuroendocrinology. 1999 Nov;24(8):813-22. doi: 10.1016/s0306-4530(99)00031-1. PMID 10581652
- [Background] Christiansen K, Knussmann R. Sex hormones and cognitive functioning in men. Neuropsychobiology. 1987;18(1):27-36. doi: 10.1159/000118389. PMID 3444523
- [Background] Morley JE, Kaiser F, Raum WJ, Perry HM 3rd, Flood JF, Jensen J, Silver AJ, Roberts E. Potentially predictive and manipulable blood serum correlates of aging in the healthy human male: progressive decreases in bioavailable testosterone, dehydroepiandrosterone sulfate, and the ratio of insulin-like growth factor 1 to growth hormone. Proc Natl Acad Sci U S A. 1997 Jul 8;94(14):7537-42. doi: 10.1073/pnas.94.14.7537. PMID 9207127
- [Background] Moffat SD, Hampson E. A curvilinear relationship between testosterone and spatial cognition in humans: possible influence of hand preference. Psychoneuroendocrinology. 1996 Apr;21(3):323-37. doi: 10.1016/0306-4530(95)00051-8. PMID 8817730
- [Background] Muller M, Aleman A, Grobbee DE, de Haan EH, van der Schouw YT. Endogenous sex hormone levels and cognitive function in aging men: is there an optimal level? Neurology. 2005 Mar 8;64(5):866-71. doi: 10.1212/01.WNL.0000153072.54068.E3. PMID 15753424
- [Background] Beauchet O. Testosterone and cognitive function: current clinical evidence of a relationship. Eur J Endocrinol. 2006 Dec;155(6):773-81. doi: 10.1530/eje.1.02306. PMID 17132744
- [Background] Stanton SJ, Liening SH, Schultheiss OC. Testosterone is positively associated with risk taking in the Iowa Gambling Task. Horm Behav. 2011 Feb;59(2):252-6. doi: 10.1016/j.yhbeh.2010.12.003. Epub 2010 Dec 15. PMID 21167166
- [Background] Apicella CL, Dreber A, Mollerstrom J. Salivary testosterone change following monetary wins and losses predicts future financial risk-taking. Psychoneuroendocrinology. 2014 Jan;39:58-64. doi: 10.1016/j.psyneuen.2013.09.025. Epub 2013 Oct 6. PMID 24275004
- [Background] Coates JM, Gurnell M, Sarnyai Z. From molecule to market: steroid hormones and financial risk-taking. Philos Trans R Soc Lond B Biol Sci. 2010 Jan 27;365(1538):331-43. doi: 10.1098/rstb.2009.0193. PMID 20026470
- [Background] Anderson RA, Martin CW, Kung AW, Everington D, Pun TC, Tan KC, Bancroft J, Sundaram K, Moo-Young AJ, Baird DT. 7Alpha-methyl-19-nortestosterone maintains sexual behavior and mood in hypogonadal men. J Clin Endocrinol Metab. 1999 Oct;84(10):3556-62. doi: 10.1210/jcem.84.10.6028. PMID 10522995
- [Background] O'Carroll R, Shapiro C, Bancroft J. Androgens, behaviour and nocturnal erection in hypogonadal men: the effects of varying the replacement dose. Clin Endocrinol (Oxf). 1985 Nov;23(5):527-38. doi: 10.1111/j.1365-2265.1985.tb01113.x. PMID 3910302
- [Background] Skakkebaek NE, Bancroft J, Davidson DW, Warner P. Androgen replacement with oral testosterone undecanoate in hypogonadal men: a double blind controlled study. Clin Endocrinol (Oxf). 1981 Jan;14(1):49-61. doi: 10.1111/j.1365-2265.1981.tb00364.x. PMID 7014044
- [Background] Salmimies P, Kockott G, Pirke KM, Vogt HJ, Schill WB. Effects of testosterone replacement on sexual behavior in hypogonadal men. Arch Sex Behav. 1982 Aug;11(4):345-53. doi: 10.1007/BF01541595. PMID 7149969
- [Background] Wang C, Swerdloff RS, Iranmanesh A, Dobs A, Snyder PJ, Cunningham G, Matsumoto AM, Weber T, Berman N; Testosterone Gel Study Group. Transdermal testosterone gel improves sexual function, mood, muscle strength, and body composition parameters in hypogonadal men. J Clin Endocrinol Metab. 2000 Aug;85(8):2839-53. doi: 10.1210/jcem.85.8.6747. PMID 10946892
- [Background] Wright ND, Bahrami B, Johnson E, Di Malta G, Rees G, Frith CD, Dolan RJ. Testosterone disrupts human collaboration by increasing egocentric choices. Proc Biol Sci. 2012 Jun 7;279(1736):2275-80. doi: 10.1098/rspb.2011.2523. Epub 2012 Feb 1. PMID 22298852
- [Background] Zak PJ, Kurzban R, Ahmadi S, Swerdloff RS, Park J, Efremidze L, Redwine K, Morgan K, Matzner W. Testosterone administration decreases generosity in the ultimatum game. PLoS One. 2009 Dec 16;4(12):e8330. doi: 10.1371/journal.pone.0008330. PMID 20016825
- [Background] Baker LA, Pearcey SM, Dabbs JM Jr. Testosterone, alcohol, and civil and rough conflict resolution strategies in lesbian couples. J Homosex. 2002;42(4):77-88. doi: 10.1300/J082v42n04_05. PMID 12243486
- [Background] Johnson RT, Breedlove SM. Human trust: testosterone raises suspicion. Proc Natl Acad Sci U S A. 2010 Jun 22;107(25):11149-50. doi: 10.1073/pnas.1005376107. Epub 2010 Jun 10. No abstract available. PMID 20538975
- [Background] van Honk J, Tuiten A, Verbaten R, van den Hout M, Koppeschaar H, Thijssen J, de Haan E. Correlations among salivary testosterone, mood, and selective attention to threat in humans. Horm Behav. 1999 Aug;36(1):17-24. doi: 10.1006/hbeh.1999.1521. PMID 10433883
- [Background] Luboshitzky R, Shen-Orr Z, Herer P. Middle-aged men secrete less testosterone at night than young healthy men. J Clin Endocrinol Metab. 2003 Jul;88(7):3160-6. doi: 10.1210/jc.2002-021920. PMID 12843160
- [Background] Penev PD. Association between sleep and morning testosterone levels in older men. Sleep. 2007 Apr;30(4):427-32. doi: 10.1093/sleep/30.4.427. PMID 17520786
- [Background] Wittert G. The relationship between sleep disorders and testosterone in men. Asian J Androl. 2014 Mar-Apr;16(2):262-5. doi: 10.4103/1008-682X.122586. PMID 24435056
- [Background] Ebstein RP, Israel S, Chew SH, Zhong S, Knafo A. Genetics of human social behavior. Neuron. 2010 Mar 25;65(6):831-44. doi: 10.1016/j.neuron.2010.02.020. PMID 20346758
- [Background] Bartels M, Van den Berg M, Sluyter F, Boomsma DI, de Geus EJ. Heritability of cortisol levels: review and simultaneous analysis of twin studies. Psychoneuroendocrinology. 2003 Feb;28(2):121-37. doi: 10.1016/s0306-4530(02)00003-3. PMID 12510008
- [Background] van Winkel R, Stefanis NC, Myin-Germeys I. Psychosocial stress and psychosis. A review of the neurobiological mechanisms and the evidence for gene-stress interaction. Schizophr Bull. 2008 Nov;34(6):1095-105. doi: 10.1093/schbul/sbn101. Epub 2008 Aug 20. PMID 18718885
- [Background] Uhart M, McCaul ME, Oswald LM, Choi L, Wand GS. GABRA6 gene polymorphism and an attenuated stress response. Mol Psychiatry. 2004 Nov;9(11):998-1006. doi: 10.1038/sj.mp.4001535. PMID 15197399
- [Background] Zhang L, Rao F, Wessel J, Kennedy BP, Rana BK, Taupenot L, Lillie EO, Cockburn M, Schork NJ, Ziegler MG, O'Connor DT. Functional allelic heterogeneity and pleiotropy of a repeat polymorphism in tyrosine hydroxylase: prediction of catecholamines and response to stress in twins. Physiol Genomics. 2004 Nov 17;19(3):277-91. doi: 10.1152/physiolgenomics.00151.2004. Epub 2004 Sep 14. PMID 15367723
- [Background] Sumithran P, Proietto J. The defence of body weight: a physiological basis for weight regain after weight loss. Clin Sci (Lond). 2013 Feb;124(4):231-41. doi: 10.1042/CS20120223. PMID 23126426
- [Background] Montani JP, Schutz Y, Dulloo AG. Dieting and weight cycling as risk factors for cardiometabolic diseases: who is really at risk? Obes Rev. 2015 Feb;16 Suppl 1:7-18. doi: 10.1111/obr.12251. PMID 25614199
- [Background] Cummings DE. Ghrelin and the short- and long-term regulation of appetite and body weight. Physiol Behav. 2006 Aug 30;89(1):71-84. doi: 10.1016/j.physbeh.2006.05.022. Epub 2006 Jul 21. PMID 16859720
- [Background] Liu J, Prudom CE, Nass R, Pezzoli SS, Oliveri MC, Johnson ML, Veldhuis P, Gordon DA, Howard AD, Witcher DR, Geysen HM, Gaylinn BD, Thorner MO. Novel ghrelin assays provide evidence for independent regulation of ghrelin acylation and secretion in healthy young men. J Clin Endocrinol Metab. 2008 May;93(5):1980-7. doi: 10.1210/jc.2007-2235. Epub 2008 Mar 18. PMID 18349056
- [Background] Asarian L, Geary N. Sex differences in the physiology of eating. Am J Physiol Regul Integr Comp Physiol. 2013 Dec;305(11):R1215-67. doi: 10.1152/ajpregu.00446.2012. Epub 2013 Jul 31. PMID 23904103
- [Background] Greenman Y, Rouach V, Limor R, Gilad S, Stern N. Testosterone is a strong correlate of ghrelin levels in men and postmenopausal women. Neuroendocrinology. 2009;89(1):79-85. doi: 10.1159/000151768. Epub 2008 Aug 28. PMID 18753737
- [Background] Pagotto U, Gambineri A, Pelusi C, Genghini S, Cacciari M, Otto B, Castaneda T, Tschop M, Pasquali R. Testosterone replacement therapy restores normal ghrelin in hypogonadal men. J Clin Endocrinol Metab. 2003 Sep;88(9):4139-43. doi: 10.1210/jc.2003-030554. PMID 12970277
- [Background] Jockenhovel F, Blum WF, Vogel E, Englaro P, Muller-Wieland D, Reinwein D, Rascher W, Krone W. Testosterone substitution normalizes elevated serum leptin levels in hypogonadal men. J Clin Endocrinol Metab. 1997 Aug;82(8):2510-3. doi: 10.1210/jcem.82.8.4174. PMID 9253326
- [Background] Lambert GP. Stress-induced gastrointestinal barrier dysfunction and its inflammatory effects. J Anim Sci. 2009 Apr;87(14 Suppl):E101-8. doi: 10.2527/jas.2008-1339. Epub 2008 Sep 12. PMID 18791134
- [Background] Teshima CW, Meddings JB. The measurement and clinical significance of intestinal permeability. Curr Gastroenterol Rep. 2008 Oct;10(5):443-9. doi: 10.1007/s11894-008-0083-y. PMID 18799118
- [Background] Baumgart DC, Dignass AU. Intestinal barrier function. Curr Opin Clin Nutr Metab Care. 2002 Nov;5(6):685-94. doi: 10.1097/00075197-200211000-00012. PMID 12394645
- [Background] Forchielli ML, Walker WA. The effect of protective nutrients on mucosal defense in the immature intestine. Acta Paediatr Suppl. 2005 Oct;94(449):74-83. doi: 10.1111/j.1651-2227.2005.tb02159.x. PMID 16214770
- [Background] McClung JP, Karl JP. Iron deficiency and obesity: the contribution of inflammation and diminished iron absorption. Nutr Rev. 2009 Feb;67(2):100-4. doi: 10.1111/j.1753-4887.2008.00145.x. PMID 19178651
- [Background] Deplancke B, Vidal O, Ganessunker D, Donovan SM, Mackie RI, Gaskins HR. Selective growth of mucolytic bacteria including Clostridium perfringens in a neonatal piglet model of total parenteral nutrition. Am J Clin Nutr. 2002 Nov;76(5):1117-25. doi: 10.1093/ajcn/76.5.1117. PMID 12399288
- [Background] Sonoyama K, Fujiwara R, Takemura N, Ogasawara T, Watanabe J, Ito H, Morita T. Response of gut microbiota to fasting and hibernation in Syrian hamsters. Appl Environ Microbiol. 2009 Oct;75(20):6451-6. doi: 10.1128/AEM.00692-09. Epub 2009 Aug 21. PMID 19700553
- [Background] Plaisancie P, Ducroc R, El Homsi M, Tsocas A, Guilmeau S, Zoghbi S, Thibaudeau O, Bado A. Luminal leptin activates mucin-secreting goblet cells in the large bowel. Am J Physiol Gastrointest Liver Physiol. 2006 Apr;290(4):G805-12. doi: 10.1152/ajpgi.00433.2005. Epub 2006 Feb 2. PMID 16455789
- [Background] Ravussin Y, Koren O, Spor A, LeDuc C, Gutman R, Stombaugh J, Knight R, Ley RE, Leibel RL. Responses of gut microbiota to diet composition and weight loss in lean and obese mice. Obesity (Silver Spring). 2012 Apr;20(4):738-47. doi: 10.1038/oby.2011.111. Epub 2011 May 19. PMID 21593810
- [Background] Braniste V, Leveque M, Buisson-Brenac C, Bueno L, Fioramonti J, Houdeau E. Oestradiol decreases colonic permeability through oestrogen receptor beta-mediated up-regulation of occludin and junctional adhesion molecule-A in epithelial cells. J Physiol. 2009 Jul 1;587(Pt 13):3317-28. doi: 10.1113/jphysiol.2009.169300. Epub 2009 May 11. PMID 19433574
- [Background] Meng J, Mostaghel EA, Vakar-Lopez F, Montgomery B, True L, Nelson PS. Testosterone regulates tight junction proteins and influences prostatic autoimmune responses. Horm Cancer. 2011 Jun;2(3):145-56. doi: 10.1007/s12672-010-0063-1. PMID 21761342
- [Background] Markle JG, Frank DN, Mortin-Toth S, Robertson CE, Feazel LM, Rolle-Kampczyk U, von Bergen M, McCoy KD, Macpherson AJ, Danska JS. Sex differences in the gut microbiome drive hormone-dependent regulation of autoimmunity. Science. 2013 Mar 1;339(6123):1084-8. doi: 10.1126/science.1233521. Epub 2013 Jan 17. PMID 23328391
- [Background] Lohman TG, Harris M, Teixeira PJ, Weiss L. Assessing body composition and changes in body composition. Another look at dual-energy X-ray absorptiometry. Ann N Y Acad Sci. 2000 May;904:45-54. doi: 10.1111/j.1749-6632.2000.tb06420.x. PMID 10865709
- [Background] Coviello AD, Kaplan B, Lakshman KM, Chen T, Singh AB, Bhasin S. Effects of graded doses of testosterone on erythropoiesis in healthy young and older men. J Clin Endocrinol Metab. 2008 Mar;93(3):914-9. doi: 10.1210/jc.2007-1692. Epub 2007 Dec 26. PMID 18160461
- [Background] Lakshman KM, Kaplan B, Travison TG, Basaria S, Knapp PE, Singh AB, LaValley MP, Mazer NA, Bhasin S. The effects of injected testosterone dose and age on the conversion of testosterone to estradiol and dihydrotestosterone in young and older men. J Clin Endocrinol Metab. 2010 Aug;95(8):3955-64. doi: 10.1210/jc.2010-0102. Epub 2010 Jun 9. PMID 20534765
- [Background] Mifflin MD, St Jeor ST, Hill LA, Scott BJ, Daugherty SA, Koh YO. A new predictive equation for resting energy expenditure in healthy individuals. Am J Clin Nutr. 1990 Feb;51(2):241-7. doi: 10.1093/ajcn/51.2.241. PMID 2305711
- [Background] Lo S, Russell JC, Taylor AW. Determination of glycogen in small tissue samples. J Appl Physiol. 1970 Feb;28(2):234-6. doi: 10.1152/jappl.1970.28.2.234. No abstract available. PMID 5413312
- [Background] Carbone JW, Margolis LM, McClung JP, Cao JJ, Murphy NE, Sauter ER, Combs GF Jr, Young AJ, Pasiakos SM. Effects of energy deficit, dietary protein, and feeding on intracellular regulators of skeletal muscle proteolysis. FASEB J. 2013 Dec;27(12):5104-11. doi: 10.1096/fj.13-239228. Epub 2013 Aug 21. PMID 23965841
- [Background] Spiering BA, Kraemer WJ, Vingren JL, Ratamess NA, Anderson JM, Armstrong LE, Nindl BC, Volek JS, Hakkinen K, Maresh CM. Elevated endogenous testosterone concentrations potentiate muscle androgen receptor responses to resistance exercise. J Steroid Biochem Mol Biol. 2009 Apr;114(3-5):195-9. doi: 10.1016/j.jsbmb.2009.02.005. Epub 2009 Feb 21. PMID 19429451
- [Background] Price JC, Holmes WE, Li KW, Floreani NA, Neese RA, Turner SM, Hellerstein MK. Measurement of human plasma proteome dynamics with (2)H(2)O and liquid chromatography tandem mass spectrometry. Anal Biochem. 2012 Jan 1;420(1):73-83. doi: 10.1016/j.ab.2011.09.007. Epub 2011 Sep 14. PMID 21964502
- [Background] Bray GA, Redman LM, de Jonge L, Covington J, Rood J, Brock C, Mancuso S, Martin CK, Smith SR. Effect of protein overfeeding on energy expenditure measured in a metabolic chamber. Am J Clin Nutr. 2015 Mar;101(3):496-505. doi: 10.3945/ajcn.114.091769. Epub 2015 Jan 14. PMID 25733634
- [Background] WEIR JB. New methods for calculating metabolic rate with special reference to protein metabolism. J Physiol. 1949 Aug;109(1-2):1-9. doi: 10.1113/jphysiol.1949.sp004363. No abstract available. PMID 15394301
- [Background] Jequier E, Acheson K, Schutz Y. Assessment of energy expenditure and fuel utilization in man. Annu Rev Nutr. 1987;7:187-208. doi: 10.1146/annurev.nu.07.070187.001155. No abstract available. PMID 3300732
- [Background] Lieberman HR, Bathalon GP, Falco CM, Kramer FM, Morgan CA 3rd, Niro P. Severe decrements in cognition function and mood induced by sleep loss, heat, dehydration, and undernutrition during simulated combat. Biol Psychiatry. 2005 Feb 15;57(4):422-9. doi: 10.1016/j.biopsych.2004.11.014. PMID 15705359
- [Background] Lieberman HR, Caruso CM, Niro PJ, Adam GE, Kellogg MD, Nindl BC, Kramer FM. A double-blind, placebo-controlled test of 2 d of calorie deprivation: effects on cognition, activity, sleep, and interstitial glucose concentrations. Am J Clin Nutr. 2008 Sep;88(3):667-76. doi: 10.1093/ajcn/88.3.667. PMID 18779282
- [Background] Butcher J, Graham J, Tellegen A, Dahlstrom W, Kaemmer B. Minnesota Multiphasic Personality Inventory-2 (MMPI-2): Manual for administration, scoring, and interpretation 2nd ed. Minneapolis, MN: University of Minnesota Press; 2001.
- [Background] Weiner IB, Greene RL. Handbook of Personality Assessment. Hoboken, NJ: Wiley; 2006.
- [Background] Spiro A, Butcher JN, Levenson RM, Aldwin CM, Bossé R. Change and stability in personality: A 5-year study of the MMPI-2 in older men. In: Butcher JN, ed. Fundamentals of MMPI-2: Research and application Minneapolis, MN: University of Minnesota Press; 2000:443-462.
- [Background] Keo-Meier CL, Herman LI, Reisner SL, Pardo ST, Sharp C, Babcock JC. Testosterone treatment and MMPI-2 improvement in transgender men: a prospective controlled study. J Consult Clin Psychol. 2015 Feb;83(1):143-56. doi: 10.1037/a0037599. Epub 2014 Aug 11. PMID 25111431
- [Background] Buss AH, Perry M. The aggression questionnaire. J Pers Soc Psychol. 1992 Sep;63(3):452-9. doi: 10.1037//0022-3514.63.3.452. PMID 1403624
- [Background] O'Connor DB, Archer J, Wu FC. Effects of testosterone on mood, aggression, and sexual behavior in young men: a double-blind, placebo-controlled, cross-over study. J Clin Endocrinol Metab. 2004 Jun;89(6):2837-45. doi: 10.1210/jc.2003-031354. PMID 15181066
- [Background] McNair DM, Lorr M, Droppleman LF. Profile of Mood States Manual. San Diego, CA: Educational and Industrial Testing Service; 1971.
- [Background] Banderet LE, Lieberman HR. Treatment with tyrosine, a neurotransmitter precursor, reduces environmental stress in humans. Brain Res Bull. 1989 Apr;22(4):759-62. doi: 10.1016/0361-9230(89)90096-8. PMID 2736402
- [Background] Lieberman HR, Bathalon GP, Falco CM, et al. The Fog of War: Documenting Cognitive Decrements Associated with the Stress of Combat. 2002.
- [Background] Lieberman HR, Falco CM, Slade SS. Carbohydrate administration during a day of sustained aerobic activity improves vigilance, as assessed by a novel ambulatory monitoring device, and mood. Am J Clin Nutr. 2002 Jul;76(1):120-7. doi: 10.1093/ajcn/76.1.120. PMID 12081825
- [Background] Lieberman HR, Tharion WJ, Shukitt-Hale B, Speckman KL, Tulley R. Effects of caffeine, sleep loss, and stress on cognitive performance and mood during U.S. Navy SEAL training. Sea-Air-Land. Psychopharmacology (Berl). 2002 Nov;164(3):250-61. doi: 10.1007/s00213-002-1217-9. Epub 2002 Sep 5. PMID 12424548
- [Background] Shukitt-Hale B, Askew EW, Lieberman HR. Effects of 30 days of undernutrition on reaction time, moods, and symptoms. Physiol Behav. 1997 Oct;62(4):783-9. doi: 10.1016/s0031-9384(97)00236-9. PMID 9284498
- [Background] Cardello AV, Schutz HG, Lesher LL, Merrill E. Development and testing of a labeled magnitude scale of perceived satiety. Appetite. 2005 Feb;44(1):1-13. doi: 10.1016/j.appet.2004.05.007. Epub 2004 Nov 13. PMID 15604029
- [Background] Lejuez CW, Read JP, Kahler CW, Richards JB, Ramsey SE, Stuart GL, Strong DR, Brown RA. Evaluation of a behavioral measure of risk taking: the Balloon Analogue Risk Task (BART). J Exp Psychol Appl. 2002 Jun;8(2):75-84. doi: 10.1037//1076-898x.8.2.75. PMID 12075692
- [Background] Burnham TC. High-testosterone men reject low ultimatum game offers. Proc Biol Sci. 2007 Sep 22;274(1623):2327-30. doi: 10.1098/rspb.2007.0546. PMID 17613451
- [Background] Baron-Cohen S, Wheelwright S, Hill J, Raste Y, Plumb I. The "Reading the Mind in the Eyes" Test revised version: a study with normal adults, and adults with Asperger syndrome or high-functioning autism. J Child Psychol Psychiatry. 2001 Feb;42(2):241-51. PMID 11280420
- [Background] Prevost M, Carrier ME, Chowne G, Zelkowitz P, Joseph L, Gold I. The Reading the Mind in the Eyes test: validation of a French version and exploration of cultural variations in a multi-ethnic city. Cogn Neuropsychiatry. 2014;19(3):189-204. doi: 10.1080/13546805.2013.823859. Epub 2013 Aug 13. PMID 23937473
- [Background] Fine BJ, Kobrick JL, Lieberman HR, Marlowe B, Riley RH, Tharion WJ. Effects of caffeine or diphenhydramine on visual vigilance. Psychopharmacology (Berl). 1994 Mar;114(2):233-8. doi: 10.1007/BF02244842. PMID 7838913
- [Background] Dinges DF, Powell JW. Microcomputer analyses of performance on a portable, simple, visual RT task during sustained operations. Vol 171985:652-655.
- [Background] Baddeley AD. A 3 min reasoning test based on grammatical transformation. Psychon Sci. 1968;10(10):341-342.
- [Background] Morgenthaler T, Alessi C, Friedman L, Owens J, Kapur V, Boehlecke B, Brown T, Chesson A Jr, Coleman J, Lee-Chiong T, Pancer J, Swick TJ; Standards of Practice Committee; American Academy of Sleep Medicine. Practice parameters for the use of actigraphy in the assessment of sleep and sleep disorders: an update for 2007. Sleep. 2007 Apr;30(4):519-29. doi: 10.1093/sleep/30.4.519. PMID 17520797
- [Background] Vartanian O, Mandel DR, Duncan M. Money or life: Behavioral and neural context effects on choice under uncertainty. Journal of Neuroscience, Psychology, and Economics. 2011;4(1):25-36.
- [Background] Lotze M, Veit R, Anders S, Birbaumer N. Evidence for a different role of the ventral and dorsal medial prefrontal cortex for social reactive aggression: An interactive fMRI study. Neuroimage. 2007 Jan 1;34(1):470-8. doi: 10.1016/j.neuroimage.2006.09.028. Epub 2006 Oct 27. PMID 17071110
- [Background] Bush G, Shin LM. The Multi-Source Interference Task: an fMRI task that reliably activates the cingulo-frontal-parietal cognitive/attention network. Nat Protoc. 2006;1(1):308-13. doi: 10.1038/nprot.2006.48. PMID 17406250
- [Background] Carter CS, Braver TS, Barch DM, Botvinick MM, Noll D, Cohen JD. Anterior cingulate cortex, error detection, and the online monitoring of performance. Science. 1998 May 1;280(5364):747-9. doi: 10.1126/science.280.5364.747. PMID 9563953
- [Background] Goetz SM, Tang L, Thomason ME, Diamond MP, Hariri AR, Carre JM. Testosterone rapidly increases neural reactivity to threat in healthy men: a novel two-step pharmacological challenge paradigm. Biol Psychiatry. 2014 Aug 15;76(4):324-31. doi: 10.1016/j.biopsych.2014.01.016. Epub 2014 Jan 29. PMID 24576686
- [Background] Blundell J, de Graaf C, Hulshof T, Jebb S, Livingstone B, Lluch A, Mela D, Salah S, Schuring E, van der Knaap H, Westerterp M. Appetite control: methodological aspects of the evaluation of foods. Obes Rev. 2010 Mar;11(3):251-70. doi: 10.1111/j.1467-789X.2010.00714.x. Epub 2010 Jan 29. PMID 20122136
- [Background] Kuczynski J, Lauber CL, Walters WA, Parfrey LW, Clemente JC, Gevers D, Knight R. Experimental and analytical tools for studying the human microbiome. Nat Rev Genet. 2011 Dec 16;13(1):47-58. doi: 10.1038/nrg3129. PMID 22179717
- [Background] Caporaso JG, Lauber CL, Walters WA, Berg-Lyons D, Huntley J, Fierer N, Owens SM, Betley J, Fraser L, Bauer M, Gormley N, Gilbert JA, Smith G, Knight R. Ultra-high-throughput microbial community analysis on the Illumina HiSeq and MiSeq platforms. ISME J. 2012 Aug;6(8):1621-4. doi: 10.1038/ismej.2012.8. Epub 2012 Mar 8. PMID 22402401
- [Background] Caporaso JG, Kuczynski J, Stombaugh J, Bittinger K, Bushman FD, Costello EK, Fierer N, Pena AG, Goodrich JK, Gordon JI, Huttley GA, Kelley ST, Knights D, Koenig JE, Ley RE, Lozupone CA, McDonald D, Muegge BD, Pirrung M, Reeder J, Sevinsky JR, Turnbaugh PJ, Walters WA, Widmann J, Yatsunenko T, Zaneveld J, Knight R. QIIME allows analysis of high-throughput community sequencing data. Nat Methods. 2010 May;7(5):335-6. doi: 10.1038/nmeth.f.303. Epub 2010 Apr 11. No abstract available. PMID 20383131
- [Background] Possemiers S, Verthe K, Uyttendaele S, Verstraete W. PCR-DGGE-based quantification of stability of the microbial community in a simulator of the human intestinal microbial ecosystem. FEMS Microbiol Ecol. 2004 Sep 1;49(3):495-507. doi: 10.1016/j.femsec.2004.05.002. PMID 19712298
- [Background] Grootjans J, Thuijls G, Verdam F, Derikx JP, Lenaerts K, Buurman WA. Non-invasive assessment of barrier integrity and function of the human gut. World J Gastrointest Surg. 2010 Mar 27;2(3):61-9. doi: 10.4240/wjgs.v2.i3.61. PMID 21160852
- [Background] Stunkard AJ, Messick S. The three-factor eating questionnaire to measure dietary restraint, disinhibition and hunger. J Psychosom Res. 1985;29(1):71-83. doi: 10.1016/0022-3999(85)90010-8. PMID 3981480
- [Background] Weiner C. Anticipate and communicate: Ethical management of incidental and secondary findings in the clinical, research, and direct-to-consumer contexts (December 2013 report of the Presidential Commission for the Study of Bioethical Issues). Am J Epidemiol. 2014 Sep 15;180(6):562-4. doi: 10.1093/aje/kwu217. Epub 2014 Aug 22. PMID 25150271
- [Derived] Margolis LM, Marlatt KL, Berryman CE, Howard EE, Murphy NE, Carrigan CT, Harris MN, Beyl RA, Ravussin E, Pasiakos SM, Rood JC. Metabolic Adaptations and Substrate Oxidation are Unaffected by Exogenous Testosterone Administration during Energy Deficit in Men. Med Sci Sports Exerc. 2023 Apr 1;55(4):661-669. doi: 10.1249/MSS.0000000000003089. Epub 2022 Nov 22. PMID 36563086
- [Derived] Vartanian O, Lam TK, Mandel DR, Ann Saint S, Navarrete G, Carmichael OT, Murray K, Pillai SR, Shankapal P, Caldwell J, Berryman CE, Karl JP, Harris M, Rood JC, Pasiakos SM, Rice E, Duncan M, Lieberman HR. Effect of exogenous testosterone in the context of energy deficit on risky choice: Behavioural and neural evidence from males. Biol Psychol. 2023 Jan;176:108468. doi: 10.1016/j.biopsycho.2022.108468. Epub 2022 Dec 5. PMID 36481265
- [Derived] Howard EE, Shankaran M, Evans WJ, Berryman CE, Margolis LM, Lieberman HR, Karl JP, Young AJ, Montano MA, Matthews MD, Bizieff A, Nyangao E, Mohammed H, Harris MN, Hellerstein MK, Rood JC, Pasiakos SM. Effects of Testosterone on Mixed-Muscle Protein Synthesis and Proteome Dynamics During Energy Deficit. J Clin Endocrinol Metab. 2022 Jul 14;107(8):e3254-e3263. doi: 10.1210/clinem/dgac295. PMID 35532889
- [Derived] Karl JP, Berryman CE, Harris MN, Lieberman HR, Gadde KM, Rood JC, Pasiakos SM. Effects of Testosterone Supplementation on Ghrelin and Appetite During and After Severe Energy Deficit in Healthy Men. J Endocr Soc. 2020 Mar 3;4(4):bvaa024. doi: 10.1210/jendso/bvaa024. eCollection 2020 Apr 1. PMID 32258956
- [Derived] Hennigar SR, Berryman CE, Harris MN, Karl JP, Lieberman HR, McClung JP, Rood JC, Pasiakos SM. Testosterone Administration During Energy Deficit Suppresses Hepcidin and Increases Iron Availability for Erythropoiesis. J Clin Endocrinol Metab. 2020 Apr 1;105(4):dgz316. doi: 10.1210/clinem/dgz316. PMID 31894236
- [Derived] Pasiakos SM, Berryman CE, Karl JP, Lieberman HR, Orr JS, Margolis LM, Caldwell JA, Young AJ, Montano MA, Evans WJ, Vartanian O, Carmichael OT, Gadde KM, Harris M, Rood JC. Physiological and psychological effects of testosterone during severe energy deficit and recovery: A study protocol for a randomized, placebo-controlled trial for Optimizing Performance for Soldiers (OPS). Contemp Clin Trials. 2017 Jul;58:47-57. doi: 10.1016/j.cct.2017.05.001. Epub 2017 May 4. PMID 28479217

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three participants discontinued the study during phase 1, prior to intervention assignment to a study arm: 1 was unable to tolerate study procedures and 2 had conflicting work/time commitments.
Groups:
- Energy Deficit: Participants randomly assigned to the control condition were subjected to exercise-induced energy expenditure resulting in a 55% energy deficit and were administered sesame oil placebo injections during phase 2 of the trial.
  Sesame Oil: 200 mg sesame oil by intramuscular injection weekly on days 15, 21, 28, and 35
- Energy Deficit + Testosterone: Participants randomly assigned to the intervention condition were subjected to exercise-induced energy expenditure resulting in a 55% energy deficit and were administered testosterone enanthate injections during phase 2 of the trial.
  testosterone enanthate: 200 mg testosterone enanthate by intramuscular injection weekly on days 15, 21, 28, and 35
Period: Overall Study
Arm/Group | Energy Deficit | Energy Deficit + Testosterone
Started | 26 | 24
Completed | 26 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Energy Deficit | Energy Deficit + Testosterone | Total
Number analyzed (Participants) | 26 | 24 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (1) | 25 (1) | 25 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 26 | 24 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic Black | 7 | 6 | 13
  Non-Hispanic White | 16 | 14 | 30
  Hispanic | 0 | 3 | 3
  Other | 3 | 1 | 4
Height [Mean (Standard Deviation); unit: centimeters] | 178 (1) | 178 (2) | 178 (7)
Weight [Mean (Standard Deviation); unit: kilograms] | 76 (2) | 81 (3) | 78 (12)
Body Mass Index [Mean (Standard Deviation); unit: kilograms per square meter] | 24 (1) | 25 (1) | 25 (3)
Systolic Blood Pressure [Mean (Standard Deviation); unit: millimeters mercury] | 117 (2) | 119 (2) | 118 (9)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: millimeters mercury] | 74 (2) | 72 (2) | 73 (7)
Total Testosterone [Mean (Standard Deviation); unit: nanograms per deciliter] | 430 (19) | 495 (27) | 461 (118)
Free Testosterone [Mean (Standard Deviation); unit: nanograms per deciliter] | 9 (1) | 10 (1) | 9.3 (2.8)
Follicle Stimulating Hormone [Mean (Standard Deviation); unit: milli-international units per milliliter] | 4 (0.4) | 3 (0.4) | 3.6 (2.1)
Estradiol [Mean (Standard Deviation); unit: picograms per milliliter] | 42 (3) | 43 (3) | 42.5 (14.2)
Sex Hormone Binding Globulin [Mean (Standard Deviation); unit: nanomoles per liter] | 32.0 (1.8) | 37.4 (3.6) | 34.5 (14.5)
Luteinizing Hormone [Mean (Standard Deviation); unit: milli-international units per milliliter] | 4.4 (2.0) | 3.7 (1.3) | 4.1 (1.7)
Insulin-like Growth Factor-1 [Mean (Standard Deviation); unit: nanograms per milliliter] | 277 (88) | 280 (72) | 278 (80)
Glucose [Mean (Standard Deviation); unit: milligrams per deciliter] | 89 (1) | 88 (1) | 88.5 (5.8)
Insulin [Mean (Standard Deviation); unit: micro-international units per milliliter] | 7.9 (7.3) | 9.7 (15.3) | 8.8 (11.8)
Cortisol [Mean (Standard Deviation); unit: micrograms per deciliter] | 14.9 (5.1) | 13.4 (3.9) | 14.2 (4.6)
Total Cholesterol [Mean (Standard Deviation); unit: milligrams per deciliter] | 168 (7) | 162 (6) | 165 (30)
High-Density Lipoprotein Cholesterol [Mean (Standard Deviation); unit: milligrams per deciliter] | 53 (2) | 57 (3) | 54.7 (11.9)
Low-Density Lipoprotein Cholesterol [Mean (Standard Deviation); unit: milligrams per deciliter] | 100 (5) | 91 (4) | 95.4 (24.4)
Triglyceride [Mean (Standard Deviation); unit: milligrams per deciliter] | 77 (9) | 72 (7) | 74.6 (40.2)
Hemoglobin [Mean (Standard Deviation); unit: grams per deciliter] | 15 (0.2) | 15 (0.2) | 15 (1)
Hematocrit [Mean (Standard Deviation); unit: percentage] | 44 (0.5) | 45 (0.5) | 44 (3)
Prostate-Specific Antigen [Mean (Standard Deviation); unit: nanograms per milliliter] | 0.65 (0.1) | 0.72 (0.1) | 0.72 (0.5)
Alanine Aminotransferase [Mean (Standard Deviation); unit: international units per liter] | 20.9 (1.6) | 23.6 (1.7) | 22.2 (8.2)
Body Mass Composition [Mean (Standard Deviation); unit: kilograms]
  Total | 76.6 (2.0) | 80.9 (2.8) | 78.7 (12.1)
  Fat-free | 56.0 (1.1) | 60.7 (2.1) | 58.2 (8.2)
  Fat | 17.4 (1.3) | 17.0 (1.4) | 17.2 (6.7)
Peak Oxygen Uptake [Mean (Standard Deviation); unit: liters per minute] | 3.4 (0.6) | 3.6 (0.8) | 3.5 (0.7)
Absolute Intake [Mean (Standard Deviation); unit: kilocalories per day]
  Energy | 2478 (950) | 2432 (777) | 2456 (863)
  Carbohydrate | 281 (114) | 258 (99) | 270 (107)
  Protein | 113 (40) | 118 (39) | 115 (39)
  Fat | 103 (49) | 106 (38) | 104 (43)
Relative Intake [Mean (Standard Deviation); unit: kilocalories/kilogram body mass/day]
  Energy | 33.1 (13.4) | 31.7 (13.4) | 32 (13)
  Carbohydrate | 3.8 (1.6) | 3.4 (1.7) | 3.6 (1.6)
  Protein | 1.5 (0.5) | 1.5 (0.6) | 1.5 (0.6)
  Fat | 1.4 (0.7) | 1.4 (0.6) | 1.4 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Body Composition at the End of Each Study Phase
Description: Height was measured using a stadiometer. Weight was measured using a calibrated digital scale. Body composition was determined using dual-energy X-ray absorptiometry. These data were used to calculate fat-free body mass, fat mass, and total body tissue mass.
Time Frame: end of each study phase: Day 11 for Phase 1, Day 39 for Phase 2, up to Day 85 for Phase 3
Measure: Least Squares Mean (95% Confidence Interval); unit: kilograms
Arm/Group | Energy Deficit | Energy Deficit + Testosterone
Number analyzed (Participants) | 26 | 24
kilograms
  Total Body Mass at end of Phase 1 | 78.3 [77.7 to 78.9] | 78.0 [77.4 to 78.7]
  Total Body Mass at end of Phase 2 | 73.3 [72.7 to 74.0] | 75.8 [75.1 to 76.5]
  Total Body Mass at end of Phase 3 | 76.5 [75.8 to 77.1] | 79.3 [78.6 to 79.9]
  Fat-free Mass at end of Phase 1 | 58.3 [57.7 to 58.9] | 57.9 [57.3 to 58.5]
  Fat-free Mass at end of Phase 2 | 58.0 [57.4 to 58.6] | 60.4 [59.8 to 61.0]
  Fat-free Mass at end of Phase 3 | 60.5 [60.0 to 61.1] | 63.1 [62.5 to 63.7]
  Fat Mass at end of Phase 1 | 16.8 [16.4 to 17.2] | 16.8 [16.3 to 17.2]
  Fat Mass at end of Phase 2 | 12.2 [11.8 to 12.6] | 12.0 [11.6 to 12.4]
  Fat Mass at end of Phase 3 | 12.8 [12.4 to 13.2] | 12.8 [12.4 to 13.2]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time of the screening visit until study completion, up to 4 months.
Groups:
- Energy Deficit: Participants randomly assigned to the control condition were subject to exercise-induced energy expenditure resulting in a 55% energy deficit and were administered sesame oil placebo injections during phase 2 of the trial.
  Sesame Oil: 200 mg sesame oil by intramuscular injection weekly on days 15, 21, 28, and 35
- Energy Deficit + Testosterone: Participants randomly assigned to the intervention condition were subject to exercise-induced energy expenditure resulting in a 55% energy deficit and were administered testosterone enanthate injections during phase 2 of the trial.
  testosterone enanthate: 200 mg testosterone enanthate by intramuscular injection weekly on days 15, 21, 28, and 35
Arm/Group | Energy Deficit | Energy Deficit + Testosterone
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/26 | 4/24
Other Adverse Events (participants affected / at risk) | 26/26 | 23/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Energy Deficit (N=26) | Energy Deficit + Testosterone (N=24)
Elevated Alanine Aminotransferase (Hepatobiliary disorders) | 0 | 2
Abnormal Lab Results (Blood and lymphatic system disorders) | 0 | 1
Biopsy Infection, Cellulitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Energy Deficit (N=26) | Energy Deficit + Testosterone (N=24)
Biopsy Pain (Surgical and medical procedures) | 20 | 19
Blister/Chafing (Skin and subcutaneous tissue disorders) | 7 | 8
Foot Pain (General disorders) | 7 | 6
Joint/Muscle Soreness (Musculoskeletal and connective tissue disorders) | 18 | 13
Gastrointestinal (Gastrointestinal disorders) | 5 | 6
Dermatological (Skin and subcutaneous tissue disorders) | 6 | 6
Insomnia (General disorders) | 6 | 9
Headache (General disorders) | 4 | 7
Allergy/Eye Irritation/Ear Pain (General disorders) | 8 | 6
Other (General disorders) | 6 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-03): https://cdn.clinicaltrials.gov/large-docs/38/NCT02734238/Prot_SAP_000.pdf